CLINICAL TRIAL: NCT01537484
Title: Multisite RCT Investigating the Efficacy of Massage in Osteoarthritis
Brief Title: Exploring Massage Benefits for Arthritis of the Knee
Acronym: EMBARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: Pro00032894; 7R01AT004623-04 (NIH)
Record Dates: First submitted 2012-02-07; First posted 2012-02-23 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2015-08

CONDITIONS: Osteoarthritis
Keywords: massage; osteoarthritis; light touch; Swedish
MeSH Terms: conditions — Osteoarthritis | interventions — Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Swedish Massage (Experimental): Swedish massage for one hour, once per week, for eight weeks. At week 10, 50% of patients will be randomized to a maintenance dose (one hour of Swedish massage every two weeks), and 50% will be randomized to Usual Care.
  Interventions: Procedure: Massage Therapy
- Light Touch Bodywork (Active Comparator): Light-touch bodywork for one hour, once per week, for eight weeks. At week 10, 50% of the patients will be randomized to a maintenance dose (one hour of light-touch massage every two weeks, and 50% will be randomized to Usual Care.
  Interventions: Procedure: Massage Therapy
- Usual Care (Other): Those initially randomized to the usual care control will be rolled into the Swedish massage intervention (one hour of Swedish massage, once/week for eight weeks) at week 25. At week 34, 50% of patients will be randomized to a maintenance dose (one hour of Swedish massage every two weeks), while 50% will be randomized back to Usual Care.
  Interventions: Procedure: Massage Therapy

INTERVENTIONS:
Procedure: Massage Therapy — Swedish Massage for 1 hour for 8 weeks, Light Touch Bodywork for 1 hours for 8 weeks.
  Other Names: Usual Care

SUMMARY:
The purpose of this study is to verify the efficacy of an 8-week course of manualized Swedish massage for reducing pain and increasing function compared to light-touch bodywork, and usual care, in 222 adults with OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

* 35 years of age or greater.
* Written confirmation of OA of the knee as provided by the participant's physician.
* Radiographically-established OA of the knee.
* Pre-randomization rating within a certain range on the Visual Analog Pain Scale (0 - 100 mm scale).
* Receiving care for diagnosed OA of the knee under the care of a board-certified primary care physician, with or without involvement of a board-certified rheumatologist.
* Patients with bilateral knee involvement will have the more severely affected knee designated as the study knee.
* American College of Rheumatology defined OA of the knee; specifically:

  a. Knee pain b. Satisfaction of at least three of the following six criteria: i. Age great than 50 years ii. Stiffness < 30 minutes iii. Crepitus iv. Bony Tenderness v. Bony enlargement vi. No palpable warmth

Exclusion Criteria:

* Presence of rheumatoid arthritis, fibromyalgia, recurrent or active pseudo gout.
* Presence of cancer or other decompensated medical conditions that limit the ability to participate fully in all interventions, assessments, and follow-up visits.
* Signs or history of kidney or liver failure.
* Presence of asthma requiring the use of corticosteroid treatment.
* Use of oral corticosteroids within the past four weeks.
* Use of intra-articular knee depo-corticosteroids with the past three months.
* Use of intra-articular hyaluronate with the past six months.
* Arthroscopic surgery of the knee within the past year.
* Significant injury to the knee within the past six months.
* Presence of a rash or open wound over the knee.
* Unable to satisfy the treatment and follow-up requirements.
* Unable to provide written informed consent.
* Currently receiving massage therapy on a regular basis (at least twice a month).
* Knee replacement of study knee (ok if the knee not being studied has been replaced).
* History of participating in the EMBARK Phase I or II studies.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Osteoarthritis of the Knee and Hip Index (WOMAC) | Baseline, 8, 16, 24, 36 and 52 weeks (Baseline, 8, 16, 24, 32, 40 and 48 for Usual Care group)
  The Index is self-administered and assesses the three dimensions of pain, disability and joint stiffness in knee and hip osteoarthritis through 24 questions. WOMAC 3.1 is available in 65 languages using either a five-point Likert scale or a 100 mm visual analog scale. The WOMAC has been subject to numerous validation studies to assess reliability and responsiveness to change in therapy, including physical forms of therapy

SECONDARY OUTCOMES:
Change in Pain: The Visual Analog Scale (VAS) | Baseline, 8, 16, 24, 36 and 52 weeks (Baseline, 8, 16, 24, 32, 40 and 48 for Usual Care group)
  Used to measure pain sensation intensity evoked by nociceptive stimuli. Subjects quickly and easily rate stimuli within the series by indicating level of pain on a 100 mm scale. Pain intensity is represented by the participant drawing a line on the scale indicative of pain experienced (0 = no pain, to 100 = worse pain imaginable). The VAS is anchored at the left by "no pain sensation" and at the right by "the most intense pain sensation imaginable."
Change in Pain: PROMIS Pain Interference Questionnaire | Baseline, 8, 16, 24, 36 and 52 weeks (Baseline, 8, 16, 24, 32, 40 and 48 for Usual Care group)
  Patient Reported Outcomes Measurement Information System (PROMIS), funded by the National Institutes of Health (NIH), is a system of highly reliable, valid, flexible, precise, and responsive assessment tools that measure patient-reported health status. The Pain Interference Questionnaire has 6 questions answered on an ordinal scale of five gradations.
Change in Joint Flexibility | Baseline, 8, 16, 24, 36 and 52 weeks (Baseline, 8, 16, 24, 32, 40 and 48 for Usual Care group)
  Joint flexibility is defined as the range of motion (ROM) allowed at the knee. The knee's ROM is measured by the number of degrees from the starting position of a segment to its position at the end of its full range of the movement. This is measured using a double-armed goniometer. A stationary arm holding a protractor is placed parallel with a stationary body segment and a movable arm moves along a moveable body segment. The pin (axis of goniometer) is placed over the joint.
Change in Physical Function | Baseline, 8, 16, 24, 36 and 52 weeks (Baseline, 8, 16, 24, 32, 40 and 48 for Usual Care group)
  Measured time in seconds to walk fifty (50) feet (15 m) on a level surface within the clinic facilities.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Perlman, MD, MPH, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Yale-Griffin Prevention Research Center, Integrative Medicine Center at Griffin Hospital, Derby, Connecticut
  - Atlantic Health System -- Atlantic Health Integrative Medicine, Morristown, New Jersey
  - Duke University Medical Center- Duke Integrative Medicine, Durham, North Carolina

REFERENCES:
- [Result] Perlman AI, Sabina A, Williams AL, Njike VY, Katz DL. Massage therapy for osteoarthritis of the knee: a randomized controlled trial. Arch Intern Med. 2006 Dec 11-25;166(22):2533-8. doi: 10.1001/archinte.166.22.2533. PMID 17159021
- [Result] Perlman AI, Ali A, Njike VY, Hom D, Davidi A, Gould-Fogerite S, Milak C, Katz DL. Massage therapy for osteoarthritis of the knee: a randomized dose-finding trial. PLoS One. 2012;7(2):e30248. doi: 10.1371/journal.pone.0030248. Epub 2012 Feb 8. PMID 22347369
- [Derived] Perlman A, Fogerite SG, Glass O, Bechard E, Ali A, Njike VY, Pieper C, Dmitrieva NO, Luciano A, Rosenberger L, Keever T, Milak C, Finkelstein EA, Mahon G, Campanile G, Cotter A, Katz DL. Efficacy and Safety of Massage for Osteoarthritis of the Knee: a Randomized Clinical Trial. J Gen Intern Med. 2019 Mar;34(3):379-386. doi: 10.1007/s11606-018-4763-5. Epub 2018 Dec 12. PMID 30543021
- See also: Duke Integrative Medicine — http://www.dukeintegrativemedicine.org